CLINICAL TRIAL: NCT07063862
Title: PSilocybin Microdose for psYCHological and Existential Distress in PALliative Care (PSYCHED-PAL): A Multi-site Phase 3 Double-blind, Placebo-controlled, Parallel-arm Clinical Trial
Brief Title: Psilocybin Microdose for Psychological and Existential Distress in Palliative Care (PSYCHED-PAL-RCT)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Responsible Party: Principal Investigator, James Downar, Senior Scientist; Head, Division of Palliative Care, University of Ottawa, Bruyère Health Research Institute.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7745629246728
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Psychological Distress
Keywords: Psychological distress; psilocybin; microdosing
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This study is a multi-site, randomized, double-blind, placebo-controlled, parallel-arm clinical trial with an optional open-label access and extension phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin Microdosing (Experimental)
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — Participants randomized to the psilocybin microdosing intervention will take 2mg (if participant weighs <55kg) or 3mg (if participant weighs ≥55 kg) of psilocybin daily on Monday, Tuesday, Thursday, and Friday for two consecutive weeks.
  Arms: Psilocybin Microdosing
Drug: Placebo — Participants randomized to the placebo intervention will take 2mg (if participant weighs <55kg) or 3mg (if participant weighs ≥55 kg) of placebo daily on Monday, Tuesday, Thursday, and Friday for two consecutive weeks.
  Arms: Placebo

SUMMARY:
About 30-50% of patients with advanced illness experience depression, anxiety, or decreased sense of purpose and autonomy. Together, these are called psychological distress. Treatment options such as medication and therapy are available; however, they do not always work and can be time-consuming and expensive. We need treatments that work well, quickly, and can be available to all patients with advanced illness who have psychological distress.

Psilocybin, a psychedelic medication (commonly called 'magic mushrooms') works well for improving psychological distress in people with cancer or chronic illness when given in high doses with specific forms of therapy. However, psilocybin has not been well-studied among people with advanced illness, and there are concerns about safety and side effects in people approaching the end of life.

However, reports on psilocybin microdosing, which involves taking small doses that do not cause hallucinations and do not require therapy, suggest that this may be effective, safer, and more acceptable for people with advanced illness. We recently completed a small study of psilocybin microdosing. Our results showed psilocybin microdose improved psychological distress in most participants with advanced illness, without serious side effects. Our next step is to do a randomized clinical trial where some patients receive psilocybin microdose and some receive placebo (a drug that contains no medicinal ingredients). By comparing these two groups, we can remove the possibility that improvements in symptoms are only because patients thought they were getting treatment.

We will enroll 120 patients from inpatient, outpatient, and community care settings across seven sites. Participants in the microdose psilocybin group will receive 2 or 3 mg of psilocybin daily, 4 days per week, for two consecutive weeks. The placebo group will receive placebo with the same treatment schedule. All participants will be offered microdose psilocybin after 2-week follow-up. If this study is successful, we have the potential to change how psychological distress is managed in patients with advanced illness.

DETAILED DESCRIPTION:
Patients with advanced illness report feeling a sense of hopelessness, loss of autonomy and relationships, and a lack of purpose in life. These feelings of psychological suffering have been described as "existential distress" and are associated with poor outcomes, including decreased medication adherence and quality of life, increased desire for hastened death and rates of suicide, and has been identified as a primary reason why individuals pursue medical assistance in dying (MAiD).

Current treatments for psychological and existential suffering have low efficacy and are challenging to use in a palliative context. Pharmacological approaches for treating psychological suffering may reduce symptoms of depression and anxiety, but evidence to support their efficacy in palliative care (PC) is underwhelming. Antidepressant and anxiolytic medications also take time to work and can cause serious side effects such as falls and confusion, which can be substantial deterrents for patients. Similarly, results from randomized controlled trials (RCTs) and meta-analyses have demonstrated psychotherapeutic interventions show limited benefit in a PC population. Further, psychotherapy can be time consuming and slow to work, which is not ideal for patients with limited life expectancy. Given the burden of psychological and existential distress among patients followed by PC providers, there is a need to develop scalable, brief, and rapidly effective therapeutic approaches to reduce this distress.

Psychedelic medications offer an innovative, safe, complementary approach to address psychological and existential suffering in patients receiving PC. Studies from the 1950's showed serotonergic hallucinogens ("psychedelics") improved depression and anxiety symptoms in cancer patients. However, legislative changes restricted the use of these medications in clinical care and research. Interest in psychedelic medications has been rekindled by two recently published RCTs that studied the use of psilocybin (a mushroom-derived 5HT2A agonist) during a single psychotherapeutic session in cancer patients with anxiety and/or depression. These trials demonstrated rapid, clinically meaningful, and long-lasting reductions in depressed mood and/or anxiety symptoms and improvements in quality of life and death acceptance. Although the exact mechanism by which psilocybin affects mood symptoms is unclear, functional MRI studies of the brain show psilocybin disrupts the functional connectivity between anterior hippocampus (involved in memory and anticipation of future events) and the default mode network (associated with anhedonia and rumination on negative themes). There is also evidence suggesting psilocybin microdosing - taking sub-hallucinogenic doses continuously over longer time periods, rather than a one-time hallucinogenic dose - can improve mood and anxiety. The effects of microdosing, however, have not been rigorously evaluated, particularly in patients with life limiting illness.

Results from recent trials are encouraging but knowledge gaps remain. First, studies to date primarily enrolled patients with localized disease who experience different distress than that of patients with advanced disease who are near the end of life. Second, it is unclear if Canadians would find psilocybin an attractive option in the context of MAiD legalization, which provides an alternative option for patients with severe psychological suffering. Third, there is no empirical research on the therapeutic effects of psilocybin microdosing, as most studies have followed macrodosing protocols. While preliminary efficacy of macrodosing has been demonstrated, there are important barriers to administering this therapy in a PC context. Previous trials had slow recruitment rates, suggesting there may be barriers related to the acceptability of psilocybin macrodosing from the perspectives of patients and families. Macrodosing requires the patient to dedicate an entire day to participating in a guided hallucinogenic experience and remain in an acute care setting where they can be closely monitored. It also requires patients to engage in preparatory sessions with monitors and a post-therapy session. In a PC context, this time commitment may not be acceptable or feasible for patients who are nearing the end of life. Macrodosing requires at least two trained moderators to guide the patient through their psychedelic experience and facilitate the pre- and post-dosing sessions. In most PC settings, it is not feasible to have clinicians dedicate two days to a single patient, thus limiting the scalability of this intervention. Anecdotally, concerns about the safety of high-dose psilocybin in the terminally ill, as well as access to psychotherapy, may also be substantial barriers in this population. Moreover, randomized trials of psychedelic medications are methodologically challenging because patients cannot be blinded to having a psychedelic experience. This "functional unblinding" was one major reason why the US FDA chose not to approve psychedelic medication for the treatment of post-traumatic stress disorder in August 2024, despite strongly positive trial results.

Psilocybin microdosing may be safer and more feasible than psilocybin macrodosing in palliative setting. Psychedelic microdosing involves taking 5-10% of a psychedelic dose of a substance such as psilocybin on a regular basis (daily or several times per week). It does not produce a psychedelic experience, nor does it involve psychotherapy, but large surveys and anecdotal reports suggest that microdosing produces substantial and sustained improvements in mood and anxiety symptoms without any important side effects. By removing the requirement for trained moderators, minimizing the time commitment required of patients, eliminating the hallucinogenic effects of the therapy, and allowing patients to receive treatment either as an inpatient or in the community, microdosing may be a more acceptable option to patients and families and allow psychedelic therapy to be scalable across various PC settings.

We have completed a phase 2 dose-finding and proof of concept study for microdosing psilocybin in people with advanced illness receiving PC. Using progressively increasing microdoses of psilocybin over a 3-week period (from 1 mg to 3 mg daily), we found that a large proportion of participants experienced dramatic improvements in their psychological distress, with minimal side effects. This effect was durable after stopping the medication but diminished after 4 weeks. Given the encouraging findings from our phase 2 study, and the potential feasibility, scalability, and safety of psilocybin microdosing for a population with few effective options, proceeding to a phase 3 placebo-controlled trial is warranted.

Objectives

Primary Objectives:

To determine the efficacy of microdose psilocybin for improving psychological distress among patients with advanced illness followed by a palliative care provider.

Secondary Objectives:

1. Assess whether microdose psilocybin improves quality of life and desire to die among patients with advanced illness followed by a palliative care provider.
2. Determine the safety of long-term (up to 1 year) use of psilocybin microdose to treat psychological distress among patients with advanced illness followed by a palliative care provider.

Open-Label Access and Extension Phase

Following the primary study 2-week follow-up completion, all participants will have the option to participate in an open-label access phase. In this phase, participants will be offered open-label psilocybin for two consecutive weeks (same dosing and schedule as the primary study). Two weeks after the access phase has been completed, all participants will have the option to participate in the open-label extension period for up to 1 year. The open-label extension will follow a three-week dosing cycle, where all participants will take psilocybin microdoses for two consecutive weeks, and then no doses on the third week, before starting the cycle again.

The open-label and open-label extension phase include safety and primary and secondary outcomes (see Outcome Measures), in line with the primary study protocol.

Sample Size

We require a sample size of 60 patients per arm (120 patients in total). This assumes a 20% loss to attrition/deterioration and 10% withdrawal (based on our phase 2 study). This sample would have 80% power to detect a change of 0.30 from 30% PGIC response (control) to 60% PGIC response (intervention) at last treatment day, corresponding to an effect size (Cohen's d) of 0.61.

Statistical Analysis

We will follow an intent-to-treat approach. We will use chi-square tests to compare the proportion of participants in the microdose psilocybin vs. placebo arm with a PGIC score of ≥5 at the last day of treatment and at 2-week follow-up, and to compare the proportion of participants who demonstrate a minimal clinically important difference (MCID) in secondary efficacy outcomes. To minimize type I error, a correction will be performed on the multiple secondary endpoint analyses.

Safety and feasibility outcomes will be analyzed using descriptive statistics with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >/=18 years of age with advanced illness under palliative care management, defined as having an estimated 2 to 12 months life expectancy (in the judgment of the palliative care provider)
2. Experiencing psychological distress, defined as a score of 7 or greater on the Depression, Anxiety, or Well-being item of the Edmonton Symptom Assessment System-revised (ESAS-r)
3. Living situation falls under one of two categories:

   1. Living in the community (i.e., receiving palliative care as an outpatient or through community home visits)
   2. Living in a chronic care inpatient facility (i.e., receiving long-term supportive care because care is unable to be provided in a community home - e.g., ALS) and have a family member who can administer the psilocybin/placebo medication to the patient
4. Ability to understand and communicate in English or French
5. For patients in community settings, patients must be able to have another individual present with them during and for 2 hours after they take their psilocybin/placebo dose for the first week of the intervention period

Exclusion Criteria:

1. Current or previously diagnosed, or first-degree relative with, psychotic or bipolar disorder
2. Previously deemed eligible for MAiD with intention to proceed with MAiD regardless of study intervention effectiveness (this criteria is meant to exclude patients who would be unlikely to complete follow-up - those considering or being assessed for MAiD will still be eligible)
3. Documented or suspected delirium in the past 3 months without a clearly defined reversible cause (e.g. opioid toxicity, infection) and resolution
4. Documented moderate or severe dementia diagnosis
5. Inability to provide first-person informed consent
6. Inability to complete assessments via telephone or video-conferencing platform
7. Severe or unstable physical symptoms based on the judgment of the palliative care provider
8. Palliative Performance Scale (PPS) <50%*
9. Cancer with known central nervous system (CNS) involvement or other CNS disease
10. Use of high-dose psychedelic substances in the past year
11. Taking lithium at any dose
12. Taking tramadol at any dose
13. Taking tapentadol at any dose
14. Taking any monoamine oxidase inhibitor at any dose [American Hospital Formulary Service (AFHS) group 28:16.04.12 or 28:36.32, including, but not limited to, moclobemide, tranylcypromine, phenelzine, selegiline, rasagiline]
15. Taking any atypical antipsychotic (aripiprazole, asenapine, brexpiprazole, clozapine, lurasidone, olanzapine, paliperidone, quetiapine, risperidone, ziprasidone)

    a. Note: patients can be included if their atypical antipsychotic is stopped or, if appropriate, substituted with haloperidol 48 hours prior to the start and for the duration of the intervention period and follow-up.
16. No enteral route of drug administration available
17. Pregnancy or lactation

    * Does not apply to the open-label access or open-label extension phases (since participants are expected to decline in overall health and function from baseline due to natural disease progression towards the end of life).

Individuals with dementia (assessed at baseline by the treating team - no formal screening of dementia will be done during the intervention or follow-up period) or delirium are excluded. While the safety and effects of psilocybin have not previously been studied in these populations, it can be reasonably assumed that hallucinogenic substances could exacerbate or lead to worsening of delirium or dementia symptoms common among people at the end of life (e.g., confusion, agitation).

The use of selective serotonin reuptake inhibitors (SSRIs) and antipsychotic medications (other than atypical antipsychotics) is a relative contraindication. For participants taking either an SSRI or an antipsychotic medication, there are several conditions for participation: (1) the palliative care provider must approve their participation in the study; (2) the SSRI/antipsychotic medication dose cannot change for the duration of the intervention trial and follow-up, and; (3) the patient must not be taking more than the maximum allowable trial dose for each SSRI.

The decision to not include SSRI and antipsychotic medications as an absolute contraindication was three-fold. Firstly, there is no empirical evidence from psilocybin microdosing literature that supports these medications as absolute contraindications. Risks related to serotonin syndrome are theoretical in nature for microdosing protocols, with no actual cases being observed. Secondly, the physician investigator team has estimated the risk to participants of rebound syndrome and associated symptoms from being taken off SSRIs and/or antipsychotics to be similar to or greater than that of serotonin syndrome. Lastly, to safely have participants stop taking SSRIs and/or antipsychotic medications, this would require a relatively long period of time (weeks to months) to taper the medication, which is not feasible for palliative care and end-of-life populations.

All trial participants must agree to not take any other psychedelic substance for the duration of the clinical trial and follow-up, and to notify the investigative team of any medication changes during intervention or follow-up. Participants must also notify the investigative team if any cannabis products are consumed during the treatment days. Participants must also agree not to take their benzodiazepine or antipsychotic medication, if applicable, within 12 hours (6 hours pre and 6 hours post) of taking their study dose. Participants must also agree not to drive or operate any heavy machinery on any treatment day after taking the drug (psilocybin or placebo) for the duration of the 2-week intervention. Lastly, for patients in the community setting, participants must agree not to take the study dose alone for the first week of the intervention; at least one individual must stay with the participant at the time they take their dose and for at least 2 hours following dose administration. This is to ensure participants are not alone in the event of a serious adverse drug reaction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Distress - Patient Global Impression of Change | Weekly (every Friday) during intervention (2 weeks) and 2-week follow-up
  Measured using the Patient Global Impression of Change (PGIC) scale (score 1-7 on one item; higher scores indicate greater positive change)

SECONDARY OUTCOMES:
Change in Psychological Distress - Anxiety, Depression, and Well-being | Baseline, weekly (every Friday) during intervention (2 weeks), and 2-week follow-up
  Measured using the Edmonton System Assessment System-revised (ESAS-r) depression, anxiety, and well-being scores (score 0-10 for each item; higher scores indicate worse symptoms)
Change in Psychological Distress - Depression and Anxiety | Baseline, weekly (every Friday) during intervention (2 weeks), and 2-week follow-up
  Measured using the Hospital Anxiety and Depression Scale (HADS)(score 0-3 on each item; higher score indicate worse anxiety/depression)
Change in Psychological Distress - Depression | Baseline, weekly (every Friday) during intervention (2 weeks), and 2-week follow-up
  Measured using the Hamilton Depression Rating Scale (HDRS)(score 0-4 on each item; higher score indicate worse depression)
Psychological Distress - Change in Existential Distress | Baseline, weekly (every Friday) during intervention (2 weeks), and 2-week follow-up
  Measured using the Demoralization Scale (DS-II) (score 0-4 on each item; higher score indicate worse demoralization)
Change in Quality of Life | Baseline, weekly (every Friday) during intervention (2 weeks), and 2-week follow-up
  Measured using the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-Les-Q-SF)(score 1-5 on each item; lower score indicate worse enjoyment and satisfaction with life)
Change in Attitude Towards Death | Baseline, weekly (every Friday) during intervention (2 weeks), and 2-week follow-up
  Measured using the Categories of Attitudes Toward Death Occurrence (CADO)(score 1-6 on one item; 4-6 indicating a wish to die)
Number of Participants with Adverse Events - Change in Blood Pressure | Baseline and daily (Monday, Tuesday, Thursday, Friday) during intervention (2 weeks)
  Proportion of participants with systolic blood pressure of > 180mmHg with symptoms or > 200mmHg (regardless of whether symptoms are present)
Number of Participants with Adverse Events - Change in Heart Rate | Baseline and daily (Monday, Tuesday, Thursday, Friday) during intervention (2 weeks)
  Proportion of participants with a resting heart rate of > 130bpm
Number of Participants with Adverse Events - Delirium | Baseline and daily (Monday, Tuesday, Thursday, Friday) during intervention (2 weeks)
  Proportion of participants who develop delirium, measured by Confusion Assessment Method (CAM) in inpatient settings or the Family Confusion Assessment Method (FAM-CAM) status in outpatient and community settings
Number of Participants with Adverse Events - Serotonin Syndrome | Weekly (every Thursday, Friday) during intervention (2 weeks)
  Proportion of participants who report a combination of tachycardia (elevated heart rate) and cognitive changes (delirium, confusion), or a tremor; diagnosed as serotonin syndrome by treating palliative care physician
Recruitment Rate | Through study completion, up 1 year
  Number of patients recruited divided by the recruitment period
Enrollment Rate | Through study completion, up to 1 year
  Number of patients enrolled divided by the number of patients approached
Intervention Completion Rate | Through study completion, up to 13 months
  Number of participants who complete the 2-week intervention divided by the number of participants enrolled
Withdrawal Rate | Through study completion, up to 14 months
  Number of participants who withdrew divided by the number of participants enrolled
Follow-up Completion Rate | Through study completion, up to 14 months
  Number of participants who complete follow-up divided by the number of participant enrolled

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - William Osler Health System, Brampton, Ontario
  - Providence Care Hospital, Kingston, Ontario
  - St. Joseph's Healthcare, London, Ontario
  - South Lake Regional Health Centre, Newmarket, Ontario
  - Bruyere Health, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe SM, Nekolaichuk C, Beaumont C, Johnson L, Myers J, Strasser F. A multicenter study comparing two numerical versions of the Edmonton Symptom Assessment System in palliative care patients. J Pain Symptom Manage. 2011 Feb;41(2):456-68. doi: 10.1016/j.jpainsymman.2010.04.020. Epub 2010 Sep 15. PMID 20832987
- [Background] Robinson S, Kissane DW, Brooker J, Hempton C, Michael N, Fischer J, Franco M, Sulistio M, Clarke DM, Ozmen M, Burney S. Refinement and revalidation of the demoralization scale: The DS-II-external validity. Cancer. 2016 Jul 15;122(14):2260-7. doi: 10.1002/cncr.30012. Epub 2016 May 12. PMID 27171544
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Johnson M, Richards W, Griffiths R. Human hallucinogen research: guidelines for safety. J Psychopharmacol. 2008 Aug;22(6):603-20. doi: 10.1177/0269881108093587. Epub 2008 Jul 1. PMID 18593734
- [Background] Anderson T, Petranker R, Christopher A, Rosenbaum D, Weissman C, Dinh-Williams LA, Hui K, Hapke E. Psychedelic microdosing benefits and challenges: an empirical codebook. Harm Reduct J. 2019 Jul 10;16(1):43. doi: 10.1186/s12954-019-0308-4. PMID 31288862
- [Background] Siegel JS, Subramanian S, Perry D, Kay B, Gordon E, Laumann T, Reneau R, Gratton C, Horan C, Metcalf N, Chacko R, Schweiger J, Wong D, Bender D, Padawer-Curry J, Raison C, Raichle M, Lenze EJ, Snyder AZ, Dosenbach NUF, Nicol G. Psilocybin desynchronizes brain networks. medRxiv [Preprint]. 2023 Aug 24:2023.08.22.23294131. doi: 10.1101/2023.08.22.23294131. PMID 37701731
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Reiche S, Hermle L, Gutwinski S, Jungaberle H, Gasser P, Majic T. Serotonergic hallucinogens in the treatment of anxiety and depression in patients suffering from a life-threatening disease: A systematic review. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Feb 2;81:1-10. doi: 10.1016/j.pnpbp.2017.09.012. Epub 2017 Sep 22. PMID 28947181
- [Background] Byock I. Taking Psychedelics Seriously. J Palliat Med. 2018 Apr;21(4):417-421. doi: 10.1089/jpm.2017.0684. Epub 2018 Jan 22. PMID 29356590
- [Background] Faller H, Schuler M, Richard M, Heckl U, Weis J, Kuffner R. Effects of psycho-oncologic interventions on emotional distress and quality of life in adult patients with cancer: systematic review and meta-analysis. J Clin Oncol. 2013 Feb 20;31(6):782-93. doi: 10.1200/JCO.2011.40.8922. Epub 2013 Jan 14. PMID 23319686
- [Background] Lo C, Hales S, Jung J, Chiu A, Panday T, Rydall A, Nissim R, Malfitano C, Petricone-Westwood D, Zimmermann C, Rodin G. Managing Cancer And Living Meaningfully (CALM): phase 2 trial of a brief individual psychotherapy for patients with advanced cancer. Palliat Med. 2014 Mar;28(3):234-42. doi: 10.1177/0269216313507757. Epub 2013 Oct 29. PMID 24170718
- [Background] Salt S, Mulvaney CA, Preston NJ. Drug therapy for symptoms associated with anxiety in adult palliative care patients. Cochrane Database Syst Rev. 2017 May 18;5(5):CD004596. doi: 10.1002/14651858.CD004596.pub3. PMID 28521070
- [Background] Kissane DW. Psychospiritual and existential distress. The challenge for palliative care. Aust Fam Physician. 2000 Nov;29(11):1022-5. PMID 11127057